CLINICAL TRIAL: NCT04602832
Title: A Randomized Controlled Trial of an Online Well-Being Intervention (The ENHANCE Program) for Improving Individuals Health and Well-Being During the COVID-19 Pandemic
Brief Title: Enduring Happiness and Continued Self-Enhancement (ENHANCE) for COVID-19
Acronym: EN-COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of British Columbia (Other)
Collaborators: University of Virginia (Other); University of Utah (Other)
Responsible Party: Principal Investigator, Lesley Lutes, Dr. Lesley Lutes, R.Psych., University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: University of British Columbia
Record Dates: First submitted 2020-10-23; First posted 2020-10-26 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-10

CONDITIONS: Well-Being
Keywords: Health and Well-Being; Positive Psychology Intervention; Online Bibliotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ENHANCE Treatment Group (Experimental): The ENHANCE program was tailored to address the current health and well-being challenges faced by individuals living in the COVID-19 pandemic. The contents of each week will focus on a new evidenced-based principle that has been shown in research to decrease negative thinking and emotions, as well as increase positive thinking, emotions, and overall physical and mental health and well-being. Each week participants will focus on the skills and methods of implementing happiness and well-being into their daily routine.
  Interventions: Other: Enduring Happiness and Continued Self-Enhancement (ENHANCE) for COVID-19
- Wait-List Control Group (No Intervention): Over the course of the study, participants will be asked to refrain from accessing the ENHANCE program materials to ensure the integrity of the research design. At the end of the study duration, participants will receive the full ENHANCE program.

INTERVENTIONS:
Other: Enduring Happiness and Continued Self-Enhancement (ENHANCE) for COVID-19 — ENHANCE is a 12-session program designed to help improve subjective well-being, especially through the challenges of a pandemic. The ENHANCE program introduces and teaches people about the evidence-based principles and skills that have been shown across decades of research to improve overall health and well-being.
  Arms: ENHANCE Treatment Group

SUMMARY:
This study is a randomized controlled trial of an online, evidenced-based intervention (the ENHANCE program) that was modified to address the health and well-being challenges of COVID-19. Eligible participants will be randomized into the ENHANCE or Wait-List Control group over a 12-week period. ENHANCE participants will be introduced, and asked to practice, 10 evidenced-based principles and skills of happiness and well-being. Participants will complete an online survey about their health and well-being at baseline, midway (or 6 weeks), post-assessment (or at the end of the 12-week study), and 3-months following the end of the study.

DETAILED DESCRIPTION:
The study is designed as a 12-week, two-armed, randomized controlled trail to assess the efficacy of a COVID-19-modified version of the Enduring Happiness and Continued Self-Enhancement (ENHANCE) program. The ENHANCE program represents a 12-week multi-construct, evidenced-based intervention for improving overall happiness and subjective well-being. The ENHANCE program was modified specifically to address the known health and well-being challenges of the COVID-19 pandemic.

Eligible participants will be randomized into either the ENHANCE program or Wait-List Control (WLC) group. ENHANCE participants will be introduced to 10 evidenced-based principles that have been shown to improve health and well-being outcomes. Participants will be further guided to systematically practice these principles in their daily lives using a small-changes approach. WLC participants will be asked to continue life a usual, and provided some additional health and well-being resources that can be accessed online to support current, ongoing distress, if needed.

Participants will be asked to complete an online survey about their emotional, social, and physical well-being at baseline (or at the start of the study), midway (or 6-weeks into the study), and at post-assessment (or at the end of the study period). At the end of the study period, all control participants will also be offered the full ENHANCE program.

Investigators expect that participants receiving the ENHANCE program will show improvements across all negative (e.g., depression, anxiety) and positive (e.g., life satisfaction, quality of life) variables from baseline to post-study. Investigators further expect there to be immediate positive health and economic outcomes linked to active participation in the ENHANCE program (versus the WLC group). Investigators believe the impacts of this research will include (a) mitigating the risk of a severe onset of mental health problems related to anxiety, depression, post-traumatic stress, and suicide, (b) increasing positive mental health and well-being, and (c) increasing physical health in participants across time.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are fluent in English and are 19 years or older.

Exclusion Criteria:

* N/A

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2020-10-14 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Beck Depression Inventory - II (BDI-II) | Baseline, Mid-assessment (6 weeks), Post-assessment (3 months), Follow-up-assessment (6 months)
  Change from baseline mood
Satisfaction With Life Scale (SWLS) | Baseline, Mid-assessment (6 weeks), Post-assessment (3 months), Follow-up-assessment (6 months)
  Change from baseline satisfaction with life
Generalized Anxiety Disorder - 7 (GAD-7) | Baseline, Mid-assessment (6 weeks), Post-assessment (3 months), Follow-up-assessment (6 months)
  Change from baseline anxiety
Patient Health Questionnaire (PHQ-9) | Baseline, Mid-assessment (6 weeks), Post-assessment (3 months), Follow-up-assessment (6 months)
  Change from baseline mood
Perceived Stress Scale (PSS) | Baseline, Mid-assessment (6 weeks), Post-assessment (3 months), Follow-up-assessment (6 months)
  Change from baseline stress
Positive and Negative Affect Scale (PANAS) | Baseline, Mid-assessment (6 weeks), Post-assessment (3 months), Follow-up-assessment (6 months)
  Change from baseline affect
Health Anxiety Inventory Short-Form (HAI-SF) | Baseline, Mid-assessment (6 weeks), Post-assessment (3 months), Follow-up-assessment (6 months)
  Change from baseline anxiety

SECONDARY OUTCOMES:
World Health Organization Quality of Life (WHOQOL - BREF) | Baseline, Mid-assessment (6 weeks), Post-assessment (3 months), Follow-up-assessment (6 months)
  Change from baseline quality of life
Meaning In Life Questionnaire (MLQ) | Baseline, Mid-assessment (6 weeks), Post-assessment (3 months), Follow-up-assessment (6 months)
  Change from baseline meaning in life
Sleep Disorder Questionnaire (SDQ) | Baseline, Mid-assessment (6 weeks), Post-assessment (3 months), Follow-up-assessment (6 months)
  Change from baseline sleep quality
Measure of Attachment Qualities (MAQ) | Baseline, Mid-assessment (6 weeks), Post-assessment (3 months), Follow-up-assessment (6 months)
  Change from baseline attachment
University of California, Los Angeles Loneliness Scale (UCLA Loneliness Scale) | Baseline, Mid-assessment (6 weeks), Post-assessment (3 months), Follow-up-assessment (6 months)
  Change from baseline loneliness
Insomnia Severity Index (ISI) | Baseline, Mid-assessment (6 weeks), Post-assessment (3 months), Follow-up-assessment (6 months)
  Change from baseline sleep quality
Paffenbarger Physical Activity Questionnaire (PPAQ) | Baseline, Mid-assessment (6 weeks), Post-assessment (3 months), Follow-up-assessment (6 months)
  Change from baseline physical activity
PTSD Checklist for the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (PCL-5) | Baseline, Mid-assessment (6 weeks), Post-assessment (3 months), Follow-up-assessment (6 months)
  Change from baseline trauma-related distress
European Quality of Life Group - 5 Dimensions - 5 Levels (EQ-5D-5L) | Baseline, Mid-assessment (6 weeks), Post-assessment (3 months), Follow-up-assessment (6 months)
  Change from baseline quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- University of British Columbia, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided
We are currently consulting with others on the grant team regarding our long-term data plan and will update with our final data sharing plan in January 2021